CLINICAL TRIAL: NCT03948451
Title: A Phase I, Open-Label Study to Characterise the Absorption, Distribution, Metabolism and Excretion Following a Single Oral Dose of [14C]AZD5718 in Healthy Male Volunteers
Brief Title: Study Evaluating the Pharmacokinetic and Mass Balance of Single Dose [14C] AZD5718 in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7550C00007
Record Dates: First submitted 2019-04-01; First posted 2019-05-14 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]AZD5718 Oral Suspension (Experimental): One 200 mg dose of [14C]AZD5718 Oral Suspension
  Interventions: Drug: [14C]AZD5718 Oral Suspension

INTERVENTIONS:
Drug: [14C]AZD5718 Oral Suspension — 200 mg dose of [14C]AZD5718 Oral Suspension
  Other Names: [14C]AZD5718

SUMMARY:
The Sponsor is developing the test medicine, AZD5718, for the potential treatment of cardiovascular disease.

The study is an open-label, single dose study involving 6 healthy male subjects. The volunteers will receive a single dose of 200 mg radiolabelled AZD5718 (14C-AZD5718 Oral Suspension) containing not more than 9.9 MBq of radiocarbon.

Volunteers will attend the clinic for 9 days (Day -1 to Day 8) to receive a single dose of the test medicine. It is planned that the volunteers will be discharged as a group once all volunteers have reached the discharge criteria. This may result in the subjects being discharged as a group prior to completion of the planned residency period. If the discharge criteria are not met by volunteers by Day 8, the individual volunteers who have not met the criteria will remain in the clinical unit for a further 48 h (until Day 10).

A follow-up call will take place 7 to 10 days after discharge to ensure the ongoing wellbeing of volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 30 to 65 years with suitable veins for cannulation or repeated venepuncture.
3. Have a body mass index of 18.5 to 35.0 kg/m2, and weigh at least 50 kg and no more than 100 kg, as measured at screening.
4. Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day).
5. Must be willing and able to communicate and participate in the whole study.
6. Must be surgically sterile or agree to adhere to the contraception requirements.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results of the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Subjects with Gilbert's syndrome or subjects with a history of cholecystectomy or gall stones.
5. Any confirmed clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the investigator.
6. Any confirmed clinically significant abnormal findings in vital signs, as judged by the investigator.
7. Any confirmed clinically significant abnormal findings in 12-lead ECG, as judged by the investigator.
8. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
9. Known or suspected history of drug or alcohol abuse within the past 2 years, as judged by the investigator.
10. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 90 days of the first administration of IMP in this study. The period of exclusion ends 90 days after the final dose. Note: subjects consented and screened, but not enrolled in this study or a previous Phase I study are not excluded.
11. Plasma donation within 1 month of screening or any blood donation/loss of more than 500 mL of blood during the 3 months prior to screening.
12. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718 or the formulation excipients. Hay fever is allowed unless it is active.
13. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission.
14. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
15. Confirmed positive screen for drugs of abuse at screening or admission to the clinical unit or positive screen for alcohol at screening or admission to the clinical unit.
16. Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Subjects should stop using these herbal medications 14 days prior to administration of [14C]AZD5718.
17. Use of any prescribed or nonprescribed medication including antacids, H2 antagonists, PPI, analgesics (other than paracetamol/acetaminophen up to 4 g/day), vitamins and minerals during the 14 days prior to administration of [14C]AZD5718 or longer if the medication has a longer half-life (see Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
18. Known or suspected history of alcohol or drug abuse or regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
19. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
20. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
21. Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (ie during the screening period) minor medical complaints that may interfere with the interpretation of the study data or are considered unlikely to comply with the study procedures, restrictions and requirements.
22. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male subjects aged 30 to 65 years
Enrollment: 6 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
The amount of AZD5718 excreted (Ae) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the amount of AZD5718 excreted (Ae)
Amount of AZD5718 excreted and expressed as a percentage of the administered dose (Fe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the amount of AZD5718 excreted and expressed as a percentage of the administered dose (Fe)
The cumulative amount of AZD5718 excreted (CumAe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD5718 excreted (CumAe)
The cumulative amount of AZD5718 excreted and expressed as a percentage of the administered dose (CumFe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD5718 excreted and expressed as a percentage of the administered dose (CumFe)
Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of urine samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of faecal samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Time to maximum concentration (tmax) for AZD5718 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of AZD5718 and total radioactivity by measuring the time to maximum concentration (tmax)
Maximum plasma concentration (cmax) for AZD5718 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of AZD5718 and total radioactivity by measuring the maximum plasma concentration (cmax)
Area under the concentration time curve to the last quantifiable concentration (AUC last) for AZD5718 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of AZD5718 and total radioactivity by measuring the concentration time curve to the last quantifiable concentration (AUC last)
Area under the concentration time curve from time zero to the last quantifiable concentration (AUC0-inf) for AZD5718 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of AZD5718 and total radioactivity by measuring the concentration time curve from time zero to the last quantifiable concentration (AUC0-inf)
Apparent terminal Elimination Half-life (t1/2,λz) for AZD5718 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of AZD5718 and total radioactivity by measuring the Elimination Half-life (t1/2,λz)
Oral clearance (CL/F) of AZD5718 | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of the oral clearance of AZD5718 by measuring the apparent oral clearance (CL/F)
Apparent Volume of Distribution (Vz/F) of AZD5718 | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of the oral PK (pharmacokinetics) of AZD5718by measuring the Apparent Volume of Distribution (Vz/F)
The amount of AZD5718 excreted (Ae) | Collection of urine and faecal samples from pre-dose until 168 hours post-dose
  Assessment of the oral PK (pharmacokinetics) of AZD5718 by measuring the amount of AZD5718 excreted (Ae)
Amount of AZD5718 excreted and expressed as a percentage of the administered dose (Fe) | Collection of urine and faecal samples from pre-dose until 168 hours post-dose
  Assessment of the oral PK (pharmacokinetics) of AZD5718 by measuring the amount of AZD5718 excreted and expressed as a percentage of the administered dose (Fe)
Renal clearance (Clr) in urine of AZD5718 | Collection of urine samples from pre-dose until 168 hours post-dose
  Assessment of the oral PK (pharmacokinetics) by measuring the renal clearance (Clr)

SECONDARY OUTCOMES:
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Blood samples collected until 168 hours post-dose
  Assessment of total radioactivity in whole blood and plasma
Number of adverse events (AE) experienced by subjects | AEs recorded from the time of informed consent until discharge from the study (168 hours post-dose)
  Safety and tolerability assessed through incidence of AE

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences Limited (indemnified by Medical Protection Society)
Locations (1):
- Research Site, Ruddington, United Kingdom